CLINICAL TRIAL: NCT03501771
Title: Effects of Acupuncture on the Radial Pressure Pulse-wave at Cunkou in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH107-REC2-022
Record Dates: First submitted 2018-03-14; First posted 2018-04-18 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Low Back Pain; Low Back Pain, Mechanical; Low Back Pain, Recurrent; Low Back Pain, Postural; Low Back Strain; Lumbago; Lumbago With Sciatica; Lumbago With Sciatica, Unspecified Side; Back Pain
Keywords: Acupuncture; Back pain; Low Back Pain; Lumbago; pulse diagnosis; radial pressure pulse
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: A single group, pre-post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture (Experimental): Acupuncture needle will be administered.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Disposable acupuncture needles will be inserted into acupoints (BL23, BL25, BL40) bilaterally for a depth of 10-30 mm

SUMMARY:
Introduction: In TCM, Pulse Diagnosis has been one of the key diagnostic components in the clinical examinations. Traditionally, the palpation of the pulse on the radial artery is subjective among the physicians. With the development of the various devices to study the radial pressure pulse wave (RPPW), these have provided a scientific and objective assessment to assist the physicians on diagnosis and treatment. The primary objective of this intervention study is to investigate the effects of Acupuncture on the RPPW at cunkou in Low Back Pain (LBP) through the pulse sphygmograph. The secondary objective is to investigate the effect of acupoint combinations on different type LBP based on TCM syndrome differentiation through the primary and secondary outcome evaluations.

Methods: A single group, pre-post intervention study in which all participants receiving the same intervention will be conducted. A total 80 participants that meet all the following criteria will be enrolled: a. at least 20 years of age of either gender; b. chief complaint being low back pain; c. diagnosis with Lumbago (ICD-9-CM 724.2) or low back pain: loin pain, low back strain and lumbago NOS (not otherwise specified) (ICD-10-CM M54.4); d. diagnosis with lumbago with sciatica (ICD-10-CM M54.5). All participants will undergo acupuncture at BI23, BI25 & Bl40 after obtaining written informed consent. Objective and subjective baseline assessments and outcome evaluations including Vital Signs, health status questionnaire, Constitution in Chinese Medicines Questionnaire (CCMQ), Oswestry Disability Index, Faces Pain Scale-Revised (FPS-R) will be performed. The primary outcome will be the assessment of RPPW at cunkou ie at Cun, Guan & Chi of both hands using Pulse Sphygmograph before and after the intervention. The secondary outcome involves evaluating low back pain using the Fingertips-to-floor test & FPS-R before and after the intervention.

Expected Outcome: The results will be analyzed and provide information which can serve as clinical evidence of the influence of acupuncture on the RPPW at cunkou. In addition, the effectiveness of the acupoint combinations on the different type of LBP based on TCM syndrome differentiation can be further investigated.

DETAILED DESCRIPTION:
Introduction: In TCM, Pulse Diagnosis has been one of the key diagnostic components in the clinical examinations. Traditionally, the palpation of the pulse on the radial artery is subjective among the physicians. With the development of the various devices to study the radial pressure pulse wave (RPPW), these have provided a scientific and objective assessment to assist the physicians on diagnosis and treatment. The primary objective of this intervention study is to investigate the effects of Acupuncture on the RPPW at cunkou in Low Back Pain (LBP) through the pulse sphygmograph. The secondary objective is to investigate the effect of acupoint combinations on different type LBP based on TCM syndrome differentiation through the primary and secondary outcome evaluations.

Methods: A single group, pre-post intervention study in which all participants receiving the same intervention will be conducted. A total 80 participants that meet all the following criteria will be enrolled: a. at least 20 years of age of either gender; b. chief complaint being low back pain; c. diagnosis with Lumbago (ICD-9-CM 724.2) or low back pain: loin pain, low back strain and lumbago NOS (not otherwise specified) (ICD-10-CM M54.4); d. diagnosis with lumbago with sciatica (ICD-10-CM M54.5). All participants will undergo acupuncture at BI23, BI25 & Bl40 after obtaining written informed consent. Objective and subjective baseline assessments and outcome evaluations including Vital Signs, health status questionnaire, Constitution in Chinese Medicines Questionnaire (CCMQ), Oswestry Disability Index, Faces Pain Scale-Revised (FPS-R) will be performed. The primary outcome will be the assessment of RPPW at cunkou ie at Cun, Guan & Chi of both hands using Pulse Sphygmograph before and after the intervention. The secondary outcome involves evaluating low back pain using the Fingertips-to-floor test & FPS-R before and after the intervention.

Expected Outcome: The results will be analyzed and provide information which can serve as clinical evidence of the influence of acupuncture on the RPPW at cunkou. In addition, the effectiveness of the acupoint combinations on the different type of LBP based on TCM syndrome differentiation can be further investigated.

Other information: The study will be conducted in China Medical University Hospital (Meide Medical Building) Acupuncture Department at No. 166, Meide St, North District, Taichung, 404. It is anticipated that there will be not more than minimum risks encountered by the participants under careful needling by qualified TCM physician with minimum 10 years of clinical experiences. Data collection shall begin as soon as the IRB approval from CMUH Research Ethics Committee is obtained as well as the required equipment is available. Expected completion date: 1 yr from IRB approval.

ELIGIBILITY:
Inclusion Criteria:

1. at least 20 years of age of either gender;
2. chief complaint being low back pain;
3. diagnosis with Lumbago (ICD-9-CM 724.2) or low back pain: loin pain, low back strain and lumbago NOS (not otherwise specified) (ICD-10-CM M54.4);
4. diagnosis with lumbago with sciatica (ICD-10-CM M54.5).

Exclusion Criteria:

* Pregnancy or lactation
* CHF, carcinomas under chemotherapy, psychological/psychiatric disorders
* Heart diseases with transplanted device such as pacemaker.
* Acute infections eg Upper Respiratory Infection (URI), Urinary Tract Infections (UTI), Acute gastroenteritis.
* Inability to undergo evaluation with the Pulse Sphygmograph
* Alcohol abuse or drug addiction
* Communication disorder
* Refusal to provide informed consent or participate in the study
* Exclusion at Project Investigator's discretion
* Participation in other clinical trials within 3 months
* Allergic to metal

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Assessment of Radial Pressure Pulse-wave at cunkou (1) | 30 min before acupuncture
  Assessment of Radial Pressure Pulse-wave at cunkou ie at Cun, Guan & Chi of both hands before and after the intervention using Pulse Sphygmograph at 30 min before acupuncture.
Assessment of Radial Pressure Pulse-wave at cunkou (2) | 10 min before acupuncture
  Assessment of Radial Pressure Pulse-wave at cunkou ie at Cun, Guan & Chi of both hands before and after the intervention using Pulse Sphygmograph at 10 min before acupuncture.
Assessment of Radial Pressure Pulse-wave at cunkou (3) | 10 min after acupuncture
  Assessment of Radial Pressure Pulse-wave at cunkou ie at Cun, Guan & Chi of both hands before and after the intervention using Pulse Sphygmograph at 10 min after acupuncture.

SECONDARY OUTCOMES:
Range of Motion: Fingertip-to-Floor (FTF) test | 1) 10 min before acupuncture; 2) 10 min after needle removal
  As LBP patients will find bending forward causes more pain and limited movement, the FTF test will be conducted which the participants will be asked to bend forward and attempt to reach the floor with their index finger. the distance between the fingertip and the floor will be measured in cm.
Faces Pain Scale - Revised (FPS-R) | 1) 20 min before acupuncture; 2) 10 min after needle removal
  The intensity of pain is measure using FPS-R developed by International Association for the Study of Pain (IASP) for pain. It is incorporated into the questionnaire with a scale of 0 (no pain) to 10 (worst pain possible)

OTHER OUTCOMES:
Vital Signs - Body temperature | 1) 30 min before acupuncture;2) 10 min before acupuncture; 3) 10 min after intervention
  Body temperature will be measured using Exergen Comfort Scanner Temporal Thermometer in degree Celsius
Vital Signs - Blood Pressure | 1) 30 min before acupuncture;2) 10 min before acupuncture; 3) 10 min after intervention
  Systolic and Diastolic blood pressure will be measured using Terumo Digital Blood Pressure Monitor ES-P401 in mmHg.
Vital Signs - Pulse rate | 1) 30 min before acupuncture;2) 10 min before acupuncture; 3) 10 min after intervention
  Pulse rate will be measured using Terumo Digital Blood Pressure Monitor ES-P401 in beats/min.
Health Status Questionnaire | 20 min before acupuncture
  Age, gender, body weight, height, health status will be obtained through the questionnaire.
Constitution in Chinese Medicine Questionnaire (CCMQ) | 20 min before acupuncture
  A questionnaire developed to assess the basic body constitution of the participants which can be categorized into 9 types based on TCM principles
Oswestry Disability Index (ODI) | 20 min before acupuncture
  The Oswestry Disability Index version 2.0 is a questionnaire developed by the Medical Research Council Group will be adopted. A Chinese 2.1 version translated by researchers in Kaohsiung Medical University already available in Taiwan will be used in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Lee, M.D.,PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided